Official Title: Implementing Inclusive Fraction Intervention Classwide

NCT Number: NCT04878757

Document Date: 04/10/2020

Informed Consent Form for Parents of Participating Students

## Vanderbilt University Institutional Review Board **Informed Consent Document for Research**

Principal Investigator: Lynn Fuchs Revision Date: April 6, 2020 Study Title: Implementing Inclusive Fraction Intervention Classwide

Institution/Hospital: Vanderbilt University

| Name of participant: | <u></u> | Age: |
|----------------------|---------|------|

Dear Parent/Guardian,

The following information is provided to inform you about the research project and your participation in it. Please read this form carefully and feel free to ask any questions you may have about this study and the information given below. You will be given an opportunity to ask questions, and your questions will be answered. Also, you will be given a copy of this consent form.

Your child does not need to be in this research study. You or your child can choose to stop being in the study at any time. If we learn something new that may affect the risks or benefits of the study, we will notify you so you can decide whether you want to remain in the study. Also, if your child's teacher changes her mind about being part of this project, we will let you know your child is no longer part of the project.

## Purpose of the study:

We are asking that your child participate in this study because we are trying to find ways to improve third- and fourth-grade students' performance on fractions. As part of this project, your child's teacher may adopt as part of her standard math program a set of classwide instructional methods that has been shown to improve fourthgrade students' fraction learning. We are interested in how students' fraction learning benefits from these instructional methods when they are used classwide. To learn about the effects of these instructional methods delivered to classwide, we need to collect information about how well students learn fractions. To collect this information, students participate in math tests we administer near the start of the school year and about 6 months later during the school year. This project may help children in two ways: by giving teachers math test information to help them plan more effective teaching programs or by helping students become stronger in math. There are no identified risks of this study. As possible inconvenience may be the time it takes your child to take the tests.

## Procedures to be followed and approximate duration of the study:

To evaluate how well the program works, we will give all children in your child's class some tests that ask them to solve math problems. Research staff on this project, who are experienced teaching children your child's age, will give the tests to all students in the class at the same time in a large group. These tests take about 60 minutes on two different days near the start of the school year. The same tests will be given about 6 months later, again in two 60-minute sessions. Also, research staff will give your child one other math test individually in a quiet location at school. The individual test takes 20 minutes.

If you provide permission for us to use the tests to evaluate the program, your child's teacher will give us the large-group tests . We will give the teacher children's scores to help her plan instruction. If you do not give permission for your child to participate in the tests, your teacher will not give us his/her tests, and we will not do the individual test. (She will keep the group tests and may choose to use them in her instructional planning.)

We are asking your permission to allow the teacher to give us your child's tests and for us to give your child the individual test. If you give permission, your child's teacher will also complete a form that tells us your child's



## Vanderbilt University Institutional Review Board Informed Consent Document for Research

Principal Investigator: Lynn Fuchs Revision Date: April 6, 2020

Study Title: Implementing Inclusive Fraction Intervention Classwide

Institution/Hospital: Vanderbilt University

date of birth, sex, race, whether he/she received English language or status or special education services, how well he/she pays attention in class, and his/her school system identification number. The school district will use this identification number to tell us whether your child's receives reduced or free lunch. Your child's teacher will also complete a form telling us your child's math scores on the February MAP tests, which the school administers to all fourth-grade children, and a form telling us the types of math intervention your child gets at school.

Teachers will audio-record all instructional lessons. This is for research staff to evaluate the extent to which teachers implement the instructional protocol as intended and to allow research staff to provide feedback to teachers regarding their instruction. Audiorecordings will be stored on a Vanderbilt University secure server. Your child's name will not be associated with the audiorecordings.

Also, if 90% of these permission forms are returned, whether or not parents agree for their child to let us use their child's tests, all children in the class will receive a free sticker or pencil. There are no plans to pay you for letting us use your child's tests.

### **Expected costs:**

There are no costs related to your participation in the study.

# Description of the discomforts, inconveniences, and/or risks that can be reasonably expected as a result of participation in this study:

We see no risk associated with your child's participation. A possible inconvenience may be the time it takes your child to take the tests. Also, we will provide test results to you, if you like. If you agree to let us use your child's tests results and would like to know the results, please complete that part of the form at the end of this letter. Then we will contact you with your child's results near the end of the school year. No one else will see your child's scores, just your child's teacher and our research staff.

## Good effects that might result from this study:

This project may provide us valuable information for developing effective instructional methods in mathematics. This project may help your child in two ways: by giving teachers math test information to help them plan more effective teaching programs and by helping your child become stronger in math.

## Study results:

We will provide your child's test results to you complete that part of the form at the end of this letter. Then we will contact you with your child's results near the end of the school year. No one else will see your child's scores, just your child's teacher and our research staff. No information or scores will be added to your child's school records and reports will not identify any individual or school. Names will be removed from tests and replaced with identification numbers.

#### **Compensation for participation:**

As explained, if 90% of these permission forms are returned, whether or not parents agree for their child to let us use their child's tests, all children in the class will receive a free sticker or pencil. There are no plans to pay you for letting us use your child's tests.



## Vanderbilt University Institutional Review Board **Informed Consent Document for Research**

Principal Investigator: Lynn Fuchs Revision Date: April 6, 2020

Study Title: Implementing Inclusive Fraction Intervention Classwide

Institution/Hospital: Vanderbilt University

## Circumstances under which the Principal Investigator may withdraw you from study participation:

If your child's teacher changes her mind about being part of this project, we will let you know your child is no longer part of the project.

## What happens if you choose to withdraw from study participation?

If you decide not to let us use your child's test scores, please understand that nothing bad will happen. Also, agreeing to let us use your child's test scores is your choice and, if you change your mind, nothing bad will happen. You can call the number provided to let us know.

#### **Contact Information:**

If you would like more information about your child's participation in this project, please call Lynn Fuchs or Amelia Malone at 615-343-4782. Also, if you have general questions about giving consent or about your child's rights as a research participant, you may call the Vanderbilt Institutional Review Board at 615-322-2918.

## **Confidentiality:**

All efforts, within reason, will be made to keep your personal information in your child's research record confidential but total confidentiality cannot be guaranteed. No information or scores will be added to your child's school records, and reports will not identify any individual or school. Names will be removed from tests and replaced with identification numbers. Research records will be stored for 1 year in locked files at Vanderbilt. Efforts will be made to keep information in your child's research record private and confidential but absolute confidentiality cannot be guaranteed. Your child's information may be shared, for example, with the Vanderbilt University Institutional Review Board. This would happen only if your child or someone else is in danger or if we are required to do so by law. Vanderbilt may also provide this project's data to other research projects not listed in this letter. If data are shared, no one will be able to figure out your child was part of this project. There are no plans to pay you for such use or transfer of information.



## Vanderbilt University Institutional Review Board **Informed Consent Document for Research**

Principal Investigator: Lynn Fuchs Revision Date: April 6, 2020

Study Title: Implementing Inclusive Fraction Intervention Classwide

Institution/Hospital: Vanderbilt University

## STATEMENT BY PERSON AGREEING TO PARTICIPATE IN THIS STUDY

I have read this informed consent document and the material contained in it has been explained to me verbally. All my questions have been answered, and I freely and voluntarily choose to participate.

| Date | Signature of Parent/Guardian |
|---|---|
| Would you like us to contact | ct you near the end of the school year with your child's test results? |
| Yes | |
| No | |
| If yes, please provide your | telephone number or U.S. Mail address: |
| Phone Number: | |
| U.S. Mail Address: | <del></del> |
| (For Vanderbilt research st | aff only: Please do not write below this line.) |
| Consent obtained by: | |
| Date | Signature |
| | Printed Name and Title |

